CLINICAL TRIAL: NCT01042028
Title: A Randomised Fase I/II Trial With Irinotecan, Cetuximab and Everolimus (ICE)Compared to Capecitabine and Oxaliplatin (CapOx) for Patients With Gemcitabin Resistant Pancreatic Cancer
Brief Title: A Randomised Trial With Irinotecan, Cetuximab and Everolimus (ICE)Compared to Capecitabine and Oxaliplatin (CapOx) for Patients With Gemcitabin Resistant Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Emergence of FOLFIRINOX and slow recruitment
Sponsor: Per Pfeiffer (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Per Pfeiffer, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ICE
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas cancer; Everolimus; Irinotecan; Cetuximab; Capecitabine; Oxaliplatin; Gemcitabine resistant pancreascancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Everolimus; Cetuximab; Irinotecan; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase II: Arm A (Experimental): Regime A-ICE On progression or unacceptable toxicity patients can cross-over from regime A to regime B
  Interventions: Drug: Everolimus, Cetuximab, Irinotecan
- Arm B (Active Comparator): Arm B: CapOx On progression or unacceptable toxicity patients can cross-over from regime B to regime A.
  Interventions: Drug: Capecitabine, Oxaliplatine

INTERVENTIONS:
Drug: Everolimus, Cetuximab, Irinotecan — Cetuximab 500 mg/m² iv biweekly Irinotecan 180 mg/m² iv biweekly Everolimus in daily MDT dosage
  Other Names: RAD001
  Arms: Phase II: Arm A
Drug: Capecitabine, Oxaliplatine — Capecitabine 1250 mg/m² bid. Oxaliplatin 70 mg/m² biweekly
  Other Names: Xeloda, Eloxatin
  Arms: Arm B

SUMMARY:
This is an open multicenter randomized phase I/II study. The main purpose with this study is to investigate dose and efficacy of a combination of Irinotecan, Cetuximab and Everolimus given biweekly to patients with local advanced or metastatic pancreatic cancer AFTER progression from 1. line treatment with Gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to study entry?
2. Patient has histologically/cytologically proven, non-resectable or metastatic, adenocarcinoma of the pancreas?
3. Progressive disease during adjuvant chemotherapy (or within 6 month after) or progressive disease during or after first line chemotherapy?
4. Former treatment with chemotherapeutic agent containing gemcitabine?
5. Is the age of the patient ≥ 18 years?
6. Is the ECOG performance status 0-1?
7. Is the absolute neutrophil count (ANC) ≥ 1.5 x 109/l?
8. Is the platelet count ≥ 75 x 109/l?
9. Is the total bilirubin ≤1.5 x UNL (upper normal limit)?
10. Patient has normal liver function? (If liver metastases are present, there is no upper limit for ALAT/SPGT/alk phosph)?
11. Creatinine clearance ≥ 30 ml/min
12. Is the patient capable of following the treatment and the plan of evaluation?

Exclusion Criteria:

1. CTC Grade 3 hyperlipidaemia (>10.34 mmol/l) in spite of treatment
2. Active former or concurrent history of malignant neoplasm, in the last 2 years?
3. Any condition or therapy which, by the investigators opinion, will expose the patient to a risk or will affect the purpose of the clinical trial?
4. Pregnant or breast feeding patient (fertile patients must use contraceptives)?
5. Infections or other serious medical conditions, which can obstruct the patient's possibility of receiving the treatment? (for instance serious heart, metabolic or lung disease)
6. Known hypersensitivity toward one or more of the parts in the treatment?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Phase I: Establish maximum tolerable (MTD) dose of ICE (Irinotecan, Cetuximab and Everolimus) | 4 months
Phase I: Determine the maximum tolerated dose (MTD) of ICE in patients with gemcitabine resistant pancreatic cancer | 4 months
Phase II: Progression-free survival as measured from inclusion to either documentation of disease progression or death | 18 months

SECONDARY OUTCOMES:
Survival All events grade 1-5 according to NCI-CTCAE in fase I All Adverse events grade 1-5 according to NCI-CTCAEW in Fase II Correlation between effect of treatment and tumourmarkers Quality of life - EORTC QLQ Time to failure of Strategy | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, MD, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Department of Oncology, Aarhus Hospital, Aarhus, Aarhus
  - Department of Oncology, Odense University Hospital, Odense, Odense